CLINICAL TRIAL: NCT03463499
Title: The Efficacy and Safety of Intravesical Hyaluronic Acid and Chondroitin Sulfate After Transurethral Resection of Hunner Lesion in Interstitial Cystitis/Bladder Pain Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-08-106
Record Dates: First submitted 2018-02-25; First posted 2018-03-13 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Hyaluronic Acid; Chondroitin Sulfates

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyaluronic Acid and Chondroitin Sulfate (Experimental): Intravesical instillation of Hyaluronic Acid and Chondroitin Sulfate After Transurethral Resection of Hunner Lesion in Interstitial Cystitis/Bladder Pain Syndrome Patients.
  Interventions: Drug: Hyaluronic Acid and Chondroitin Sulfate

INTERVENTIONS:
Drug: Hyaluronic Acid and Chondroitin Sulfate — Intravesical instillation of Hyaluronic Acid and Chondroitin Sulfate After Transurethral Resection of Hunner Lesion in Interstitial Cystitis/Bladder Pain Syndrome Patients.

SUMMARY:
The efficacy and safety of intravesical hyaluronic acid and chondroitin sulfate after transurethral resection of Hunner lesion in interstitial cystitis/bladder pain syndrome patients. To analyze the number and timing of recurrence based on a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 20 yrs or greater
2. Patients diagnosed with Hunner lesion in IC(interstitial cystitis)/BPS(Bladder Pain Syndrome) and who is scheduled to undergo transurethral resection
3. Symptom persisted more than 6 months
4. Pain VAS ≥4

Exclusion Criteria:

1. History of augmentation cystoplasty or previous transurethral coagulation/resection due to IC/BPS
2. Child-bearing potential, pregnant or nursing women.
3. Hematuria exceeds 1+ in the urinary dipstick (dipstick) examination.
4. Urinary tract infection during run-in periods.
5. Genitourinary tuberculosis or bladder,urethral and prostate cancer
6. Recurrent urinary tract infection
7. History of hysterectomy,mid-urethral sling,pelvic organ prolapse repair,vaginal delivery or Cesarean section,prostate operation or treatment etc within 6months.
8. Neurologic disease history of cerebral infarction,multiple sclerosis or parkinsonism etc.-
9. Using a indwelling catheter or execution of intermittent self catheterization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
change in recurrence rate in Hyaluronic Acid and Chondroitin Sulfate instillation group after transurethral resection treatment | Every 3 months for 2 years

SECONDARY OUTCOMES:
changes in mean number of daytime frequency episodes | Every 3 months for 2 years
changes in mean number of nocturia episodes | Every 3 months for 2 years
changes in mean number of urgency episodes | Every 3 months for 2 years
Change score of O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) | Every 3 months for 2 years
Change score of Pelvic Pain and Urgency/Frequency Patient Symptom Scale(PUF) | Every 3 months for 2 years
Score of Global Response Assessment (GRA) | Every 3 months for 2 years
Patient Global Assessment | at the end of the treatment(2 years)
Occurrence of adverse event | Every 3 months for 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No